CLINICAL TRIAL: NCT06062875
Title: Effects of TNF Blockade on Human BPH/LUTS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Endeavor Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Alexander Glaser, M.D.; Clinical Assistant Professor University of Chicago Pritzker School of Medicine, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EH22-232; R01DK135516 (NIH)
Record Dates: First submitted 2023-08-29; First posted 2023-10-02 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Benign Prostatic Hyperplasia (BPH)
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Adalimumab

STUDY DESIGN:
Intervention Model Description: The purpose of this study is to investigate whether an anti-inflammatory drug commonly used for a range of autoimmune diseases may be useful to provide symptomatic relief, prostate shrinkage, and/or decrease prostatic inflammation in patients with benign prostatic hyperplasia (BPH), sometimes described as prostatic enlargement.
Masking Description: Patients will then be randomized in a double-blind fashion to receive adalimumab 40 mg every 2 weeks or placebo injection (saline) every 2 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- adalimumab (Active Comparator): adalimumab 40 mg every 2 weeks
  Interventions: Drug: Adalimumab
- Placebo (No Intervention): placebo injection (saline) every 2 weeks.

INTERVENTIONS:
Drug: Adalimumab — Adalimumab will be delivered subcutaneously (under the skin) at a dose of 40mg every 2 weeks for a total of 6 doses.
  Other Names: Placebo will be administered subcutaneously every 2 weeks, for a total of 6 injections.
  Arms: adalimumab

SUMMARY:
Specific Aim 1. To evaluate the efficacy of TNF antagonist action in BPH/LUTS Specific Aim 2. Define the consequences of TNF antagonist therapy on prostate tissue Specific Aim 3. Identify genetic predictors to stratify patients with differential response to TNF-antagonist therapy.

DETAILED DESCRIPTION:
The purpose of this study is to investigate whether an anti-inflammatory drug commonly used for a range of autoimmune diseases may be useful to provide symptomatic relief, prostate shrinkage, and/or decrease prostatic inflammation in patients with benign prostatic hyperplasia (BPH), sometimes described as prostatic enlargement.

BPH includes a significant amount of inflammation. Prior studies show that there are common links between autoimmune diseases, inflammation, and BPH. TNF-antagonists such as adalimumab are anti-inflammatory drugs commonly prescribed to treat autoimmune diseases. NorthShore researchers, including Drs. Glaser, Hayward, and Helfand, showed that these drugs reduced the incidence of BPH in patients with autoimmune diseases.

In this study, the investigators will study the TNF-antagonist adalimumab in patients with BPH who do not have autoimmune diseases. Adalimumab used in this study is investigational because it is not approved by the FDA for BPH. However, adalimumab is an approved, widely-prescribed, and commonly used drug utilized in a variety of conditions including rheumatoid arthritis, juvenile idiopathic arthritis, psoriatic arthritis, ankylosing spondylitis, Crohn's disease, ulcerative colitis, plaque psoriasis, hidradenitis suppurativa, and uveitis. It has a well-studied side effect profile and was approved for use by the FDA in 2008. The purpose of this study is to determine whether adalimumab is an effective way to reduce symptoms and/or prostatic inflammation in BPH patients without autoimmune diseases. If this research is successful it may open up a new method of therapy for patients with BPH and associated symptoms.

This study will include a total of 70 subjects. Of those subjects, all 70 will be from NorthShore University HealthSystem ("NorthShore").

ELIGIBILITY:
Inclusion Criteria:

* Male sex
* Age 45-80 years
* Diagnosed by physician with BPH
* Prostate volume ≥ 60mL
* IPSS ≥ 8
* Able and willing to complete questionnaires
* Able and willing to provide informed consent
* Able to read, write, and speak in English
* No prior treatment with TNF inhibitor (adalimumab, etanercept, infliximab, certolizumab, golimumab)
* No plans to move from study area in the next 6 months

Deferral Criteria:

* Microscopic hematuria without appropriate workup per AUA/Society of Urodynamics, Female Pelvic Medicine & Urogenital Reconstruction (SUFU) Guidelines
* Positive urine culture

Exclusion Criteria:

* Female sex or intersex
* Age < 45 or > 80 years
* Being a prisoner or detainee
* Urinary retention with need for catheterization
* Gross hematuria
* Contraindication to treatment with adalimumab (e.g., presence of sepsis or active infection, active tuberculosis, Hepatitis B infection, invasive fungal infection, lymphoma, leukemia or other active malignancy, congestive heart failure, significant hematologic abnormality, allergy to adalimumab or its components, anti-drug antibodies, congestive heart failure)
* Diagnosis of autoimmune disease (rheumatoid arthritis, plaque psoriasis, ulcerative colitis, Crohn's disease, hidradenitis suppurativa, spondyloarthritis)
* Interstitial cystitis
* Pelvic or endoscopic genitourinary surgery within the preceding 6 months (not including diagnostic cystoscopy)
* History of lower urinary tract or pelvic malignancy including prostate cancer; history of pelvic radiation therapy
* Ongoing symptomatic urethral stricture
* Current chemotherapy or other cancer therapy
* Severe neurological or psychiatric disorder that would prevent study participation (e.g., bipolar disorder, psychotic disorder, Alzheimer's Disease)
* Current moderate or severe substance use disorder

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men 45-80 years old with BPH
Enrollment: 70 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
International Prostate Symptom Score | The past 30 days
  The IPSS is a self-report measure used to assess urinary urgency, frequency, and voiding symptoms, and includes one disease-specific quality of life (QoL) question. IPSS scores ranges from 0 to 35, with higher scores indicating more severe urinary symptoms, and QoL ranges from 0 (delighted) to 6 (terrible).
Safety as measured by Clavien-Dindo grading system | Through study completion (Week 24)
  Frequency and severity of treatment related adverse events will be reported using the Clavien-Dindo severity grading system.

SECONDARY OUTCOMES:
LURN Symptom Index 29 (LURN SI-29) | The past 7 days
  This is a multidimensional 29-item questionnaire that assesses different lower urinary tract symptoms as well as single item about global bother.
The Patient-Reported Outcomes Measurement Information System (PROMIS-29) Profile v2.1 | The past 7 days
  The PROMIS-29 Profile is a 29-item instrument that combines short assessments of eight core constructs of health-related quality of life (HRQoL): physical function (PF), sleep disturbance (SD), pain interference (PI) and pain intensity (PIN), fatigue (FA), anxiety (AN), depression (DE) and ability to participate in social roles and activities (SRAA).
Patient Global Impression of Improvement (PGI-I) | Through study completion (Week 24)
  This is a single item that captures how much better or worse the person's condition is relative to when they began treatment. Scale ranges from "Very much worse" to "Very much better".
3-Day Voiding Diary | Recorded on three separate days
  The diary records the patient's daily fluid intake, frequency of urination throughout the day and night, instances of leakage, and the quantity of lost urine. Analyzing these findings against the standard criteria for regular bladder function could reveal potential issues and help confirm a diagnosis. The definition of normal benchmarks takes into account factors like age, gender, as well as various internal and external variables including fluid consumption and its nature.
Change in maximum flow rate (uroflowmetry) | Through study completion (Week 24)
  Uroflowmetry is a diagnostic test that measures the rate and pattern of urine flow during voiding to assess the functioning of the urinary tract. Changes in maximum flow rate (Qmax) will be compared.
Change in PVR (post-void residual) | Through study completion (Week 24)
  Bladder scanner to measure post-void residual
Change in prostate volume | 12 weeks
  Prostate volume as calculated by MRI prostate before and after adalimumab/placebo treatment
Change in systemic markers of inflammation (ESR, CRP) | 12 weeks
  Blood test for systemic markers of inflammation (erythrocyte sedimentation rate [ESR] and c-reactive protein [CRP]) before and after adalimumab/placebo treatment

OTHER OUTCOMES:
Cellular consequences of adalimumab therapy on prostate tissue | Through study completion (Week 24)
  We hypothesize that TNF-antagonist treatment will de-repress apoptosis, suppress proliferative pathways, and modify the immune cell profile in the prostate. In this aim we will employ flow cytometry and scRNA-seq analysis with pathway imputation, supplemented with immunohistochemistry and bulk RNA-seq, to characterize these changes at a cellular and tissue level.
Genetic predictors to stratify patients with differential response to adalimumab | Through study completion (Week 24)
  We hypothesize that genetic variants in 1) genes involved in the TNF-antagonist targeted pathways, 2) susceptibility to chronic inflammation, and 3) susceptibility to BPH influence the effectiveness of the therapy

CONTACTS AND LOCATIONS:
Overall Officials: Simon W Hayward, Ph.D., Principal Investigator — Endeavor Health; Alexander P Glaser, M.D., Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Glenview, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Reporting of results in ClinicalTrials.gov
Supporting Information: CSR
Time Frame: 08/10/2023 to June 1,2028
Access Criteria: Reporting of results in ClinicalTrials.gov Sharing of study data per NIH policies

REFERENCES:
- [Background] Vickman RE, Aaron-Brooks L, Zhang R, Lanman NA, Lapin B, Gil V, Greenberg M, Sasaki T, Cresswell GM, Broman MM, Paez JS, Petkewicz J, Talaty P, Helfand BT, Glaser AP, Wang CH, Franco OE, Ratliff TL, Nastiuk KL, Crawford SE, Hayward SW. TNF is a potential therapeutic target to suppress prostatic inflammation and hyperplasia in autoimmune disease. Nat Commun. 2022 Apr 19;13(1):2133. doi: 10.1038/s41467-022-29719-1. PMID 35440548
- [Background] Kramer G, Mitteregger D, Marberger M. Is benign prostatic hyperplasia (BPH) an immune inflammatory disease? Eur Urol. 2007 May;51(5):1202-16. doi: 10.1016/j.eururo.2006.12.011. Epub 2006 Dec 11. PMID 17182170
- [Background] Glaser AP, Mansfield S, Smith AR, Helfand BT, Lai HH, Sarma A, Yang CC, Taddeo M, Clemens JQ, Cameron AP, Flynn KE, Andreev V, Fraser MO, Erickson BA, Kirkali Z, Griffith JW; LURN Study Group. Impact of Sleep Disturbance, Physical Function, Depression and Anxiety on Male Lower Urinary Tract Symptoms: Results from the Symptoms of Lower Urinary Tract Dysfunction Research Network (LURN). J Urol. 2022 Jul;208(1):155-163. doi: 10.1097/JU.0000000000002493. Epub 2022 Feb 25. PMID 35212573
- [Background] Liu G, Andreev VP, Helmuth ME, Yang CC, Lai HH, Smith AR, Wiseman JB, Merion RM, Erickson BA, Cella D, Griffith JW, Gore JL, DeLancey JOL, Kirkali Z; LURN Study Group. Symptom Based Clustering of Men in the LURN Observational Cohort Study. J Urol. 2019 Dec;202(6):1230-1239. doi: 10.1097/JU.0000000000000354. Epub 2019 May 23. PMID 31120372
- [Background] Helfand BT, Smith AR, Lai HH, Yang CC, Gore JL, Erickson BA, Kreder KJ, Cameron AP, Weinfurt KP, Griffith JW, Lentz A, Talaty P, Andreev VP, Kirkali Z; LURN. Prevalence and Characteristics of Urinary Incontinence in a Treatment Seeking Male Prospective Cohort: Results from the LURN Study. J Urol. 2018 Aug;200(2):397-404. doi: 10.1016/j.juro.2018.02.075. Epub 2018 Mar 1. PMID 29477718
- [Background] Helfand BT, Glaser AP, Kasraeian A, Sterious S, Talaty P, Alcantara M, Alcantara KM, Higgins A, Ghiraldi E, Elterman D. Men with lower urinary tract symptoms secondary to BPH undergoing Aquablation with very large prostates (> 150 mL). Can J Urol. 2021 Dec;28(6):10884-10888. PMID 34895392
- [Background] Helfand BT, Kasraeian A, Sterious S, Glaser AP, Talaty P, Alcantara M, Alcantara KM, Higgins A, Ghiraldi E, Elterman DS. How I do it: Aquablation in very large prostates (> 150 mL). Can J Urol. 2022 Apr;29(2):11111-11115. PMID 35429430
- [Background] McConnell JD, Bruskewitz R, Walsh P, Andriole G, Lieber M, Holtgrewe HL, Albertsen P, Roehrborn CG, Nickel JC, Wang DZ, Taylor AM, Waldstreicher J. The effect of finasteride on the risk of acute urinary retention and the need for surgical treatment among men with benign prostatic hyperplasia. Finasteride Long-Term Efficacy and Safety Study Group. N Engl J Med. 1998 Feb 26;338(9):557-63. doi: 10.1056/NEJM199802263380901. PMID 9475762
- [Background] McConnell JD, Roehrborn CG, Bautista OM, Andriole GL Jr, Dixon CM, Kusek JW, Lepor H, McVary KT, Nyberg LM Jr, Clarke HS, Crawford ED, Diokno A, Foley JP, Foster HE, Jacobs SC, Kaplan SA, Kreder KJ, Lieber MM, Lucia MS, Miller GJ, Menon M, Milam DF, Ramsdell JW, Schenkman NS, Slawin KM, Smith JA; Medical Therapy of Prostatic Symptoms (MTOPS) Research Group. The long-term effect of doxazosin, finasteride, and combination therapy on the clinical progression of benign prostatic hyperplasia. N Engl J Med. 2003 Dec 18;349(25):2387-98. doi: 10.1056/NEJMoa030656. PMID 14681504
- [Background] Roehrborn CG, Bruskewitz R, Nickel JC, McConnell JD, Saltzman B, Gittelman MC, Malek GH, Gottesman JE, Suryawanshi S, Drisko J, Meehan A, Waldstreicher J; Proscar Long-Term Efficacy and Safety Study Group. Sustained decrease in incidence of acute urinary retention and surgery with finasteride for 6 years in men with benign prostatic hyperplasia. J Urol. 2004 Mar;171(3):1194-8. doi: 10.1097/01.ju.0000112918.74410.94. PMID 14767299
- [Background] Setia SA, Smith J, Cendo D, Yoder J, Gorin MA, Allaway MJ, Vourganti S. Outcomes of freehand transperineal prostate biopsy with omission of antibiotic prophylaxis. BJU Int. 2022 Jul;130(1):54-61. doi: 10.1111/bju.15590. Epub 2021 Dec 23. PMID 34491606
- [Background] Lightner DJ, Wymer K, Sanchez J, Kavoussi L. Best Practice Statement on Urologic Procedures and Antimicrobial Prophylaxis. J Urol. 2020 Feb;203(2):351-356. doi: 10.1097/JU.0000000000000509. Epub 2019 Aug 23. PMID 31441676
- [Background] He J, Guo Z, Huang Y, Wang Z, Huang L, Li B, Bai Z, Wang S, Xiang S, Gu C, Pan J. Comparisons of efficacy and complications between transrectal and transperineal prostate biopsy with or without antibiotic prophylaxis. Urol Oncol. 2022 May;40(5):191.e9-191.e14. doi: 10.1016/j.urolonc.2022.01.004. Epub 2022 Feb 12. PMID 35168882
- [Background] Ahmed Ali U, Martin ST, Rao AD, Kiran RP. Impact of preoperative immunosuppressive agents on postoperative outcomes in Crohn's disease. Dis Colon Rectum. 2014 May;57(5):663-74. doi: 10.1097/DCR.0000000000000099. PMID 24819109
- [Background] Quaresma AB, Yamamoto T, Kotze PG. Biologics and surgical outcomes in Crohn's disease: is there a direct relationship? Therap Adv Gastroenterol. 2020 Jul 16;13:1756284820931738. doi: 10.1177/1756284820931738. eCollection 2020. PMID 32728389
- [Background] Hyman NH, Cheifetz AS. PUCCINI: Safety of Anti-TNF in the Perioperative Setting. Gastroenterology. 2022 Jul;163(1):44-46. doi: 10.1053/j.gastro.2022.04.050. Epub 2022 May 4. No abstract available. PMID 35525321
- [Background] Cohen BL, Fleshner P, Kane SV, Herfarth HH, Palekar N, Farraye FA, Leighton JA, Katz JA, Cohen RD, Gerich ME, Cross RK, Higgins PDR, Tinsley A, Glover S, Siegel CA, Bohl JL, Iskandar H, Ji J, Hu L, Sands BE. Prospective Cohort Study to Investigate the Safety of Preoperative Tumor Necrosis Factor Inhibitor Exposure in Patients With Inflammatory Bowel Disease Undergoing Intra-abdominal Surgery. Gastroenterology. 2022 Jul;163(1):204-221. doi: 10.1053/j.gastro.2022.03.057. Epub 2022 Apr 10. PMID 35413359
- [Background] Bechara FG, Podda M, Prens EP, Horvath B, Giamarellos-Bourboulis EJ, Alavi A, Szepietowski JC, Kirby J, Geng Z, Jean C, Jemec GBE, Zouboulis CC. Efficacy and Safety of Adalimumab in Conjunction With Surgery in Moderate to Severe Hidradenitis Suppurativa: The SHARPS Randomized Clinical Trial. JAMA Surg. 2021 Nov 1;156(11):1001-1009. doi: 10.1001/jamasurg.2021.3655. PMID 34406349
- See also: HIGHLIGHTS OF PRESCRIBING INFORMATION — https://www.accessdata.fda.gov/drugsatfda_docs/label/2011/125057s0276lbl.pdf